CLINICAL TRIAL: NCT01033734
Title: An Open Label, Prospective, Pharmacokinetic/Pharmacodynamic and Safety Evaluation of Intravenous Oseltamivir (Tamiflu) in the Treatment of Children 1 to 12 Years of Age With Influenza Infection
Brief Title: A Study of Intravenous Tamiflu (Oseltamivir) in Children With Influenza
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP25139
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: oseltamivir [Tamiflu]

INTERVENTIONS:
Drug: oseltamivir [Tamiflu] — 5-day course (10 doses), intravenous administration, may be switched to oral administration at the discretion of the investigator; up to 5 additional days of treatment possible.

SUMMARY:
This open-label study will assess the pharmacokinetics/pharmacodynamics and safety of intravenous (iv) Tamiflu (oseltamivir) in 3 cohorts of children, aged 6-12, 3-5 and 1-2 years, with influenza infection. Patients will receive iv Tamiflu therapy for 5 days (10 doses). For patients whose conditions no longer merit continued iv dosing, therapy may be switched to oral Tamiflu to complete their prescribed course of treatment. If medically necessary, iv or oral therapy with Tamiflu may be continued for up to 5 additional days. Anticipated time on study treatment is 5 to 10 days.

ELIGIBILITY:
Inclusion Criteria:

* children, 1-12 years of age
* diagnosis of influenza
* duration of influenza symptoms </=96 hours prior to first dose of study drug

Exclusion Criteria:

* evidence of severe hepatic decompensation
* patients taking probenecid within 1 week prior to first dose of study drug

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (35):
- United States (33):
  - Los Angeles, California
  - Oakland, California
  - Aurora, Colorado
  - Wilmington, Delaware
  - Jacksonville, Florida
  - Chicago, Illinois
  - South Bend, Indiana
  - Wichita, Kansas
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Duluth, Minnesota
  - Omaha, Nebraska
  - Morristown, New Jersey
  - Brooklyn, New York
  - New York, New York
  - Stony Brook, New York
  - Syracuse, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Tyrone, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Houston, Texas
  - Richmond, Virginia
  - Madison, Wisconsin
- Petah Tikva, Israel
- Beirut, Lebanon

REFERENCES:
- [Derived] Munoz FM, Anderson EJ, Deville JG, Clinch B, Kamal MA. Pharmacokinetics and safety of intravenous oseltamivir in infants and children in open-label studies. Int J Clin Pharmacol Ther. 2015 Jul;53(7):531-40. doi: 10.5414/CP202307. PMID 26042486

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2836 participants were prescreened, of which, 2828 failed evaluation. The most common reasons for screen failure included: negative influenza diagnosis, not meeting the age criterion, ability to tolerate/absorb oral medication, and an inability to comply with the study procedures.
Groups:
- Oseltamivir: Overall: Participants received oseltamivir (Tamiflu) twice daily (every 12 hours) intravenously (IV) over 5 or 6 days for a total of 10 doses. The oseltamivir doses were based on participant's body weight. Participants with body weight less than or equal to (≤) 23 kilogram (kg) received 3 milligrams per kilogram (mg/kg); participants with body weight more than (>) 23 kg to 40 kg received 2.5 mg/kg; and participants with body weight >40 kg received 100 milligrams (mg). For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
Period: Overall Study
Arm/Group | Oseltamivir: Overall
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All-participants population included all participants who were enrolled in the study.
Groups:
- Oseltamivir: Overall: Participants received oseltamivir (Tamiflu) twice daily IV over 5 or 6 days for a total of 10 doses. The oseltamivir doses were based on participant's body weight. Participants with body weight ≤23 kg received 3 mg/kg; participants with body weight ˃23 kg to 40 kg received 2.5 mg/kg; and participants with body weight ˃40 kg received 100 mg. For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
Arm/Group | Oseltamivir: Overall
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.8 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to Last Measurable Plasma Concentration (AUClast) of Oseltamivir and Oseltamivir Carboxylate on Day 1
Time Frame: Day 1: 15 minutes pre-infusion start, 1, 2, 3, 4, 6, 8, 12 hours post start of infusion.
Population: Pharmacokinetic (PK) population included all treated participants who had at least one blood sample evaluable for drug concentration level. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter (h*ng/mL)
Groups:
- Oseltamivir: 6 to 12 Years: Participants aged 6 to 12 years received oseltamivir twice daily (every 12 hours) IV over 5 or 6 days for a total of 10 doses. The oseltamivir doses were based on participant's body weight. Participants with body weight less than or equal to 23 kg received 3 mg/kg; participants with body weight more than 23 kg to 40 kg received 2.5 mg/kg; and participants with body weight more than 40 kg received 100 mg. For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
- Oseltamivir: 3 to 5 Years: Participants aged 3 to 5 years received oseltamivir twice daily (every 12 hours) IV over 5 or 6 days for a total of 10 doses. The oseltamivir doses were based on participant's body weight. Participants with body weight less than or equal to 23 kg received 3 mg/kg; participants with body weight more than 23 kg to 40 kg received 2.5 mg/kg; and participants with body weight more than 40 kg received 100 mg. For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
- Oseltamivir: 1 to 2 Years: Participants aged 1 to 2 Years received oseltamivir twice daily (every 12 hours) IV over 5 or 6 days for a total of 10 doses. The oseltamivir doses were based on participant's body weight. Participants with body weight less than or equal to 23 kg received 3 mg/kg; participants with body weight more than 23 kg to 40 kg received 2.5 mg/kg; and participants with body weight more than 40 kg received 100 mg. For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
Arm/Group | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 1 | 3 | 0
hour*nanogram/milliliter (h*ng/mL)
  Oseltamivir | 829 | 1460 (46.3) |
  Oseltamivir Carboxylate | 1700 | 4550 (61.1) |

2. Primary Outcome: AUClast of Oseltamivir and Oseltamivir Carboxylate on Day 2
Time Frame: Day 2: 15 minutes pre-infusion start, 2, 4, 8 hours after start of infusion
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 0 | 1 | 1
h*ng/mL
  Oseltamivir |  | 1070 | 1920
  Oseltamivir Carboxylate |  | 5970 | 6760

3. Primary Outcome: AUClast of Oseltamivir and Oseltamivir Carboxylate on Day 3
Time Frame: Day 3 (with or after fifth dose): 15 minutes pre-infusion start, 2, 4, 8 hours after start of infusion
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 1 | 0 | 0
hr*ng/mL
  Oseltamivir | 943 |  |
  Oseltamivir Carboxylate | 2000 |  |

4. Primary Outcome: AUClast of Oseltamivir and Oseltamivir Carboxylate on Day 4
Time Frame: Day 4: 15 minutes pre-infusion start, 2, 4, 8 hours after start of infusion
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 0 | 1 | 0
hr*ng/mL
  Oseltamivir |  | 2480 |
  Oseltamivir Carboxylate |  | 3800 |

5. Primary Outcome: AUClast of Oseltamivir and Oseltamivir Carboxylate on Day 5
Time Frame: Day 5: 15 minutes pre-infusion start, 2, 4, 8 hours after start of infusion
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 1 | 0 | 0
hr*ng/mL
  Oseltamivir | 1010 |  |
  Oseltamivir Carboxylate | 2820 |  |

6. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Oseltamivir and Oseltamivir Carboxylate Day 1
Time Frame: Day 1: 15 minutes pre-infusion start, 1, 2, 3, 4, 6, 8, 12 hours post start of infusion
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 1 | 3 | 0
nanograms/milliliter (ng/mL)
  Oseltamivir | 360 | 753 (36.9) |
  Oseltamivir Carboxylate | 311 | 499 (55.1) |

7. Primary Outcome: Cmax of Oseltamivir and Oseltamivir Carboxylate Day 2
Time Frame: Day 2: 15 minutes pre-infusion start, 2, 4, 8 hours after start of infusion
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 0 | 1 | 1
ng/mL
  Oseltamivir |  | 500 | 1270
  Oseltamivir Carboxylate |  | 663 | 725

8. Primary Outcome: Cmax of Oseltamivir and Oseltamivir Carboxylate Day 3
Time Frame: Day 3 (with or after fifth dose): 15 minutes pre-infusion start, 2, 4, 8 hours after start of infusion
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 1 | 0 | 0
ng/mL
  Oseltamivir | 404 |  |
  Oseltamivir Carboxylate | 237 |  |

9. Primary Outcome: Cmax of Oseltamivir and Oseltamivir Carboxylate Day 4
Time Frame: Day 4: 15 minutes pre-infusion start, 2, 4, 8 hours after start of infusion
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 0 | 1 | 0
ng/mL
  Oseltamivir |  | 915 |
  Oseltamivir Carboxylate |  | 549 |

10. Primary Outcome: Cmax of Oseltamivir and Oseltamivir Carboxylate Day 5
Time Frame: Day 5: 15 minutes pre-infusion start, 2, 4, 8 hours after start of infusion
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 1 | 0 | 0
ng/mL
  Oseltamivir | 403 |  |
  Oseltamivir Carboxylate | 408 |  |

11. Secondary Outcome: Time to the Maximum Observed Plasma Concentration (Tmax) of Oseltamivir and Oseltamivir Carboxylate
Time Frame: Day 1: 15 minutes pre-infusion start, 1, 2, 3, 4, 6, 8, 12 hours post start of infusion; Day 2, 3 (with or after fifth dose), 4 or 5: 15 minutes pre-infusion start, 2, 4, 8 hours after start of infusion
Population: PK population. Number of participants analyzed = participants who were evaluable for this outcome, n = number of participants evaluable for specified categories.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 1 | 3 | 1
hours
  Day 1: Oseltamivir (n = 1, 3, 0) | 2.00 | 1.26 (41.7) | NA (NA) — Data not available as no participant was evaluable
  Day 1: Oseltamivir Carboxylate (n = 1, 3, 0) | 4.00 | 4.61 (53.3) | NA (NA) — Data not available as no participant was evaluable
  Day 2: Oseltamivir (n = 0, 1, 1) | NA (NA) — Data not available as no participant was evaluable | 2.00 (NA) — Data not available as no participant was evaluable | 1.00
  Day 2: Oseltamivir Carboxylate (n = 0, 1, 1) | NA (NA) — Data not available as no participant was evaluable | 4.62 (NA) — Data not available as no participant was evaluable | 6.00
  Day 3: Oseltamivir (n = 1, 0, 0) | 1.05 | NA (NA) — Data not available as no participant was evaluable | NA (NA) — Data not available as no participant was evaluable
  Day 3: Oseltamivir Carboxylate (n = 1, 0, 0) | 3.05 | NA (NA) — Data not available as no participant was evaluable | NA (NA) — Data not available as no participant was evaluable
  Day 4: Oseltamivir (n = 0, 1, 0) | NA (NA) — Data not available as no participant was evaluable | 2.50 (NA) — Standard deviation not applicable as only 1 participant was evaluable | NA (NA) — Data not available as no participant was evaluable
  Day 4: Oseltamivir Carboxylate (n = 0, 1, 0) | NA (NA) — Data not available as no participant was evaluable | 8.05 (NA) — Standard deviation not applicable as only 1 participant was evaluable | NA (NA) — Data not available as no participant was evaluable
  Day 5: Oseltamivir (n = 1, 0, 0) | 2.00 | NA (NA) — Data not available as no participant was evaluable | NA (NA) — Data not available as no participant was evaluable
  Day 5: Oseltamivir Carboxylate (n = 1, 0, 0) | 4.08 | NA (NA) — Data not available as no participant was evaluable | NA (NA) — Data not available as no participant was evaluable

12. Secondary Outcome: Last Measurable Plasma Concentration (Clast) of Oseltamivir and Oseltamivir Carboxylate
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 1 | 3 | 1
ng/mL
  Day 1: Oseltamivir (n = 1, 3, 0) | 4.40 | 2.41 (80.6) | NA (NA) — Data not available as no participant was evaluable.
  Day 1: Oseltamivir Carboxylate (n = 1, 3, 0) | 237 | 308 (74.4) | NA (NA) — Data not available as no participant was evaluable.
  Day 2: Oseltamivir (n = 0, 2, 1) | NA (NA) — Data not available as no participant was evaluable. | 25.2 (1704911.2) | 4.76
  Day 2: Oseltamivir Carboxylate (n = 0, 2, 1) | NA (NA) — Data not available as no participant was evaluable. | 319 (0.44) | 484
  Day 3: Oseltamivir (n = 1, 0, 0) | 2.60 | NA (NA) — Data not available as no participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Day 3: Oseltamivir Carboxylate (n = 1, 0, 0) | 149 | NA (NA) — Data not available as no participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Day 4: Oseltamivir (n = 0, 1, 0) | NA (NA) — Data not available as no participant was evaluable. | 25.1 (NA) — Standard deviation not applicable as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Day 4: Oseltamivir Carboxylate (n = 0, 1, 0) | NA (NA) — Data not available as no participant was evaluable. | 549 (NA) — Standard deviation not applicable as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Day 5: Oseltamivir (n = 1, 0, 0) | 15.1 | NA (NA) — Data not available as no participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Day 5: Oseltamivir Carboxylate (n = 1, 0, 0) | 339 | NA (NA) — Data not available as no participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.

13. Secondary Outcome: Time of the Last Measurable Plasma Concentration (Tlast) of Oseltamivir and Oseltamivir Carboxylate
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 1 | 3 | 1
hours
  Day 1: Oseltamivir (n = 1, 3, 0) | 7.42 | 10.50 (23.4) | NA (NA) — Data not available as no participant was evaluable.
  Day 1: Oseltamivir Carboxylate (n = 1, 3, 0) | 7.42 | 11.98 (0.2) | NA (NA) — Data not available as no participant was evaluable.
  Day 2: Oseltamivir (n = 0, 2, 1) | NA (NA) — Data not available as no participant was evaluable. | 3.50 (448.5) | 12.00
  Day 2: Oseltamivir Carboxylate (n = 0, 2, 1) | NA (NA) — Data not available as no participant was evaluable. | 3.50 (448.47) | 12.00
  Day 3: Oseltamivir (n = 1, 0, 0) | 10.13 | NA (NA) — Data not available as no participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Day 3: Oseltamivir Carboxylate (n = 1, 0, 0) | 10.13 | NA (NA) — Data not available as no participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Day 4: Oseltamivir (n = 0, 1, 0) | NA (NA) — Data not available as no participant was evaluable. | 8.05 (NA) — Standard deviation not applicable as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Day 4: Oseltamivir Carboxylate (n = 0, 1, 0) | NA (NA) — Data not available as no participant was evaluable. | 8.05 (NA) — Standard deviation not applicable as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Day 5: Oseltamivir (n = 1, 0, 0) | 7.92 | NA (NA) — Data not available as no participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Day 5: Oseltamivir Carboxylate (n = 1, 0, 0) | 7.92 | NA (NA) — Data not available as no participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.

14. Secondary Outcome: Elimination Rate Constant (ke) of Oseltamivir and Oseltamivir Carboxylate
Time Frame: as for outcome 11
Population: Data not available as no participant was evaluable for specified time-points.
Groups:
- Oseltamivir: Overall: Participants received oseltamivir (Tamiflu) twice daily IV over 5 or 6 days for a total of 10 doses. The oseltamivir doses were based on participant's body weight. Participants with body weight <= 23 kg received 3 mg/kg; participants with body weight ˃23 kg to 40 kg received 2.5 mg/kg; and participants with body weight ˃40 kg received 100 mg. For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
Arm/Group | Oseltamivir: Overall
Number analyzed (Participants) | 0

15. Secondary Outcome: Total Clearance of Drug (CL) of Oseltamivir and Oseltamivir Carboxylate
Time Frame: as for outcome 11
Population: Data not available as no participant was evaluable for specified time-points.
Arm/Group | Oseltamivir: Overall
Number analyzed (Participants) | 0

16. Secondary Outcome: Volume of Distribution (V) of Oseltamivir and Oseltamivir Carboxylate
Time Frame: as for outcome 11
Population: Data not collected because of changes in planned analysis, due to early study termination.
Arm/Group | Oseltamivir: Overall
Number analyzed (Participants) | 0

17. Secondary Outcome: Participants With Greater Than or Equal to (>=) 5-Fold Change in Neuraminidase Inhibition (NAI) Assay 50 Percent (%) Inhibitory Concentration (IC50) Values
Description: IC50 was defined as the concentration that causes 50% inhibition of viral activity. IC50 values were calculated using NAI assay. The 5-fold change was calculated as either >=5 times change in the NAI IC50 visit value from the Reference value at a visit, >=5 times change in the NAI IC50 Visit value from the Baseline value.
Time Frame: Baseline, Day 1, 6 and 30
Population: Safety population included all participants who received at least one dose of IV study medication and had a safety assessment performed after initiation of treatment. Here, number of participants analyzed = participants evaluable for this outcome measure, and n = participants evaluable for specified time-point, for each arm, respectively.
Measure: Number; unit: Participants
Groups:
- Oseltamivir: 6 to 12 Years: Participants aged 6 to 12 years received oseltamivir twice daily IV over 5 or 6 days for a total of 10 doses. The oseltamivir doses were based on participant's body weight. Participants with body weight <=23 kg received 3 mg/kg; participants with body weight ˃23 kg to 40 kg received 2.5 mg/kg; and participants with body weight >40 kg received 100 mg. For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
- Oseltamivir: 3 to 5 Years: Participants aged 3 to 5 years received oseltamivir twice daily IV over 5 or 6 days for a total of 10 doses. The oseltamivir doses were based on participant's body weight. Participants with body weight <=23 kg received 3 mg/kg; participants with body weight ˃23 kg to 40 kg received 2.5 mg/kg; and participants with body weight ˃40 kg received 100 mg. For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
- Oseltamivir: 1 to 2 Years: Participants aged 1 to 2 Years received oseltamivir twice daily IV over 5 or 6 days for a total of 10 doses. The oseltamivir doses were based on participant's body weight. Participants with body weight <=23 kg received 3 mg/kg; participants with body weight ˃23 kg to 40 kg received 2.5 mg/kg; and participants with body weight ˃40 kg received 100 mg. For participants who did not receive all 10 doses IV, treatment could be completed with oral oseltamivir suspension (twice daily). If medically necessary, participants were allowed to receive an additional 10 doses of IV or oral oseltamivir after the initial 10 doses.
Arm/Group | Oseltamivir: Overall | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Number analyzed (Participants) | 6 | 2 | 3 | 1
Participants
  Day 1 (n=6, 2, 3, 1) | 1 | 0 | 1 | 0
  Day 6 (n=1, 0, 1, 0) | 1 | NA — Data not available as no participant was evaluable in this arm for specified time-point. | 1 | NA — Data not available as no participant was evaluable in this arm for specified time-point.
  Day 30 (n=1, 1, 0, 0) | 0 | 0 | NA — Data not available as no participant was evaluable in this arm for specified time-point. | NA — Data not available as no participant was evaluable in this arm for specified time-point.

ADVERSE EVENTS:
Time Frame: Up to 30 days
Arm/Group | Oseltamivir: Overall | Oseltamivir: 6 to 12 Years | Oseltamivir: 3 to 5 Years | Oseltamivir: 1 to 2 Years
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/2 | 1/5 | 0/1
Other Adverse Events (participants affected / at risk) | 5/8 | 0/2 | 4/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oseltamivir: Overall (N=8) | Oseltamivir: 6 to 12 Years (N=2) | Oseltamivir: 3 to 5 Years (N=5) | Oseltamivir: 1 to 2 Years (N=1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oseltamivir: Overall (N=8) | Oseltamivir: 6 to 12 Years (N=2) | Oseltamivir: 3 to 5 Years (N=5) | Oseltamivir: 1 to 2 Years (N=1)
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter Site Erosion (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Device Expulsion (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Drug Withdrawal Syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infusion Site Erythema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Body Temperature Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain of Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Low number of participants enrolled in the study at the time that the study was terminated limits conclusions that can be derived from the study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.